CLINICAL TRIAL: NCT02041078
Title: Randomized Phase 2 Study of Intra Versus Extrahepatic Division of Right Hepatic Vein During Rightsided Hemihepatectomy
Brief Title: Intra Versus Extrahepatic Division of Right Hepatic Vein During Rightsided Hemihepatectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karolinska University Hospital (Other)
Collaborators: Jansson, Anders, M.D. (Individual); Bengt Isaksson (Unknown)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2011/563-31/2; 2011/563-31/2 (Other: Ethic committee at Karolinska Institutet Stockholm Sweden)
Record Dates: First submitted 2013-10-09; First posted 2014-01-20 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Reduction of Peroperative Blood Loss During Liver Resection
Keywords: Liver surgery; Blood loss; CUSA; Hepatic transection
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extrahepatic vein division (Placebo Comparator): Conventional right sided hemihepatectomy with division of the liver parenchyma with CUSA.
  Interventions: Procedure: Extrahepatic vein division
- Intrahepatic vein division (Experimental): Conventional right sided hemihepatectomy with division of the liver parenchyma with CUSA and intrahepatic division of the right hepatic vein.
  Interventions: Procedure: Intrahepatic division of the right hepatic vein.

INTERVENTIONS:
Procedure: Intrahepatic division of the right hepatic vein. — Ligation and division of the entrance of the right hepatic vein into the suprarenal cava vein are done at the end of transection of the liver parenchyma with CUSA.
  Arms: Intrahepatic vein division
Procedure: Extrahepatic vein division — Standard surgical procedure with extrahepatic ligation/division of the right hepatic vein prior to parenchymal division with CUSA.
  Arms: Extrahepatic vein division

SUMMARY:
Intrahepatic division of the hepatic vein is associated with less blood loss than extrahepatic dissection and division of the right hepatic vein.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic lesion amenable to right sided hemihepatectomy.

Exclusion Criteria:

* Hepatic lesions not suitable for a anatomical right sided hemihepatectomy.
* Unfit for surgery
* Unwillingness to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Intraoperative bloodloss | Intraoperative time (in minutes) for the division of the liver parenchyma

SECONDARY OUTCOMES:
Operation time, postoperative complication rate | Total time in minutes spent in theater, in hospital stay in days (on an average less than 30 days), total complication rate during hospital stay (on an average less than 30 days), surgical complications during in hospital stay (on an average<30days).
postoperative complication rate | in hospital stay in days (on an average <30 days), total complication rate during hospital stay (on an average <30 days), surgical complications during in hospital stay (on an average <30 days).

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lundell, Professor, Principal Investigator — Gastrocentrum Karolinska University Hospital Huddinge, 141 86 Stockholm
Locations (1):
- Department of Surgery Gastrocentrum Karolinska Univeristy Hospital, Stockholm, Sweden